CLINICAL TRIAL: NCT03001479
Title: Extensively Hydrolyzed Liquid Human Milk Fortifier Versus Liquid Human Milk Fortifier With Supplemental Liquid Protein
Brief Title: Noninferiority Trial of Liquid Human Milk Fortifier (HMF) Hydrolyzed Protein Versus Liquid HMF With Supplemental Liquid Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Catherine Cibulskis, MD, Assistant Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27563
Record Dates: First submitted 2016-09-20; First posted 2016-12-23 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Human Milk; Premature Birth of Newborn
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard: Liquid HMF and liquid protein (No Intervention): This is our standard breast milk fortification in our NICU. One packet (5 mL) of Similac Human Milk Fortifier Concentrated Liquid is added to breast milk feedings when infants reach 100 ml/kg/day. A second packet is added the next day (10 mL total), to make 24 kcal/oz. After infants reach full feedings (160 ml/kg/d), 3 ml/kg of Similac Liquid Protein Fortifier is added (0.5 g/kg protein). This is increased to 6 ml/kg (1 g/kg protein) the next day.
- Intervention: HMF Hydrolyzed Protein Concentrated Liquid (Experimental): One packet (5 mL) of Similac Human Milk Fortifier Hydrolyzed Protein Concentrated Liquid is added to breast milk feedings when infants reach 100 ml/kg/day. A second packet is added the next day (10 mL total), to make 24 kcal/oz. Feedings then continue to be advanced to full volume (160 ml/kg/d).
  Interventions: Dietary Supplement: Similac Human Milk Fortifier Hydrolyzed Protein Concentrated Liquid

INTERVENTIONS:
Dietary Supplement: Similac Human Milk Fortifier Hydrolyzed Protein Concentrated Liquid — HMF with additional hydrolyzed protein
  Arms: Intervention: HMF Hydrolyzed Protein Concentrated Liquid

SUMMARY:
Breast milk is readily accepted as the ideal source of nutrition for almost all infants, including premature or very low birth weight infants. However, these high-risk infants require the addition of fortifiers to their milk in order to achieve sufficient levels of calories, vitamins, and minerals for adequate growth. We are currently using a liquid human milk fortifier which does not provide sufficient protein intake, requiring addition of a liquid protein supplement. A new product has been released which provides sufficient protein in the liquid HMF, without the acidification seen in previous products.

This is a prospective, randomized noninferiority study comparing the safety and efficacy of the new HMF with additional protein to our current standard of adding additional protein supplementation on top of the HMF.

DETAILED DESCRIPTION:
All infants admitted to the Neonatal Intensive Care Unit (NICU) at Cardinal Glennon at gestational age <32 weeks and birthweight <1500g, and whose mothers intend to use breast milk (maternal or donor) will be approached for study participation. Infants can be enrolled at any point up until their feedings become fortified, typically around the 8th day of life.

Eligible infants whose parents consent for participation will be randomized to one of the two study regimens. Sealed envelopes containing the subject treatment group will be prepared from randomization schedules that are computer-generated using a pseudorandom permuted blocks algorithm. Multiples will be randomized together to the same treatment group. The randomization will be block stratified by birth weight (500-1000g and 1001-1500g). Infants will have laboratory values to follow for signs of metabolic acidosis and nutritional status. These labs (BMP, Magnesium, Phosphorous, Alkaline Phosphatase, and prealbumin) will be drawn on study days 1, 15, and 30. Total blood volume for these labs is approximately 1.4 mL, and may be obtained by venipuncture or heel stick. These labs are monitored for nutritional sufficiency in very low birth weight infants already, the only change will be the timing that the labs are obtained.

Infants will remain on their designated HMF until one of 3 different time points: 1) Infant does not tolerate HMF and must be taken off, 2) Infant is no longer receiving breastmilk and is transitioned to a premature formula, or 3) Infant is getting ready to go home and HMF is removed from the feedings.

Hospitalization data will be collected on the infants until they are either discharged from the NICU or until they reach 36 weeks corrected gestational age, whichever occurs first. Data collected will include: birthweight, gestational age, gender, antenatal steroids, APGARs, days of parenteral nutrition, day enteral feedings were initiated, daily enteral volume intake, daily caloric and protein intake, day of HMF and/or liquid protein initiation. Lab data will be recorded as noted above. Growth data will be recorded by daily weights and weekly head circumferences and lengths. Intolerance will be assessed by incidence of feeding intolerance, nil per os (NPO) time, change in diet due to intolerance, incidence of metabolic acidosis, incidence of necrotizing enterocolitis, incidence of spontaneous intestinal perforation, cause of death, and length of hospital stay. Data on NICU complications, including late onset sepsis, retinopathy of prematurity, intraventricular hemorrhage, bronchopulmonary dysplasia, and use of postnatal steroids (which can affect growth) will also be recorded.

Neurodevelopmental data will be collected on the infants from their first Bayley evaluation in the Nursery Follow-up clinic, usually performed at 15-18 months of age. We will record cognitive, language, and motor scores. We will also collect information on therapy services received, and incidence of blindness or deafness.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight, premature infants admitted to the NICU at Cardinal Glennon
* <32 weeks gestational age and birthweight <1500 grams
* receiving maternal or donor breast milk

Exclusion Criteria:

* Infants with an estimated gestational age >32 weeks OR birthweight >1500 grams
* Infants who die before fortification of feedings
* Infants receiving formula
* Infants that did not receive feedings with HMF
* Infants transferred to another hospital prior to discharge

Max Age: 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Weight gain, short term | 30 days
  (grams) in first 30 days on HMF
Length, short term | 30 days
  (cm) in first 30 days on HMF
Head circumference, short term | 30 days
  (cm) in first 30 days on HMF

SECONDARY OUTCOMES:
Weight gain, long term | 36 weeks gestational age or time of hospital discharge
  Weight (grams) at 36 weeks corrected gestational age or time of hospital discharge, whichever is first
Length, long term | 36 weeks gestational age or time of hospital discharge
  Length (cm) at 36 weeks corrected gestational age or time of hospital discharge, whichever is first
Head circumference, long term | 36 weeks gestational age or time of hospital discharge
  Head circumference (cm) at 36 weeks corrected gestational age or time of hospital discharge, whichever is first
feeding intolerance | 30 days
  Signs of feeding intolerance, including loose stools, emesis, metabolic acidosis, necrotizing enterocolitis. Presence or absence of symptoms.
neurodevelopmental outcomes | 18 months corrected gestational age
  Bayley Scales of Infant Development III at 18 months of corrected gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Catherine C Cibulskis, MD, Principal Investigator — St. Louis University
Locations (1):
- Cardinal Glennon Children's Medical Center, St Louis, Missouri, United States